CLINICAL TRIAL: NCT05503524
Title: Extensive Clinical Trial Experiences of Multiple Sclerosis Patients To Determine Trial Attributes Affecting Completion Rates For Specific Demographic Groups
Brief Title: Finding Patterns In Clinical Study Experiences of Multiple Sclerosis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 98852353
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Sclerosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participation in medical trials usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This study will admit a wide range of data on the clinical trial experience of Multiple Sclerosis patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future Multiple Sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of Multiple Sclerosis
* Patient has self-identified as planning to enroll in an interventional clinical trial for Multiple Sclerosis
* Patient is at least 18 years of age

Exclusion Criteria:

* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form
* No diagnosis of Multiple Sclerosis confirmed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Sclerosis patients who are actively considering involvement in an interventional clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a Multiple Sclerosis Clinical Trial | 3 months
Number of patients who remain in Multiple Sclerosis clinical trial until completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] He A, Merkel B, Brown JWL, Zhovits Ryerson L, Kister I, Malpas CB, Sharmin S, Horakova D, Kubala Havrdova E, Spelman T, Izquierdo G, Eichau S, Trojano M, Lugaresi A, Hupperts R, Sola P, Ferraro D, Lycke J, Grand'Maison F, Prat A, Girard M, Duquette P, Larochelle C, Svenningsson A, Petersen T, Grammond P, Granella F, Van Pesch V, Bergamaschi R, McGuigan C, Coles A, Hillert J, Piehl F, Butzkueven H, Kalincik T; MSBase study group. Timing of high-efficacy therapy for multiple sclerosis: a retrospective observational cohort study. Lancet Neurol. 2020 Apr;19(4):307-316. doi: 10.1016/S1474-4422(20)30067-3. Epub 2020 Mar 18. PMID 32199096
- [Background] Lublin FD, Reingold SC, Cohen JA, Cutter GR, Sorensen PS, Thompson AJ, Wolinsky JS, Balcer LJ, Banwell B, Barkhof F, Bebo B Jr, Calabresi PA, Clanet M, Comi G, Fox RJ, Freedman MS, Goodman AD, Inglese M, Kappos L, Kieseier BC, Lincoln JA, Lubetzki C, Miller AE, Montalban X, O'Connor PW, Petkau J, Pozzilli C, Rudick RA, Sormani MP, Stuve O, Waubant E, Polman CH. Defining the clinical course of multiple sclerosis: the 2013 revisions. Neurology. 2014 Jul 15;83(3):278-86. doi: 10.1212/WNL.0000000000000560. Epub 2014 May 28. PMID 24871874
- [Background] Belbasis L, Bellou V, Evangelou E, Ioannidis JP, Tzoulaki I. Environmental risk factors and multiple sclerosis: an umbrella review of systematic reviews and meta-analyses. Lancet Neurol. 2015 Mar;14(3):263-73. doi: 10.1016/S1474-4422(14)70267-4. Epub 2015 Feb 4. PMID 25662901

DOCUMENTS (1):
  • Informed Consent Form (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT05503524/ICF_000.pdf